CLINICAL TRIAL: NCT04857359
Title: Phase 2b/3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Dipraglurant (ADX48621) for the Treatment of Dyskinesia in Patients With Parkinson's Disease Receiving Levodopa-based Therapy
Brief Title: Dipraglurant (ADX48621) for the Treatment of Patients With Parkinson's Disease Receiving Levodopa-based Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated prior to completing enrollment goals due to COVID-related difficulties in recruiting patients
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX48621-301
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Dyskinesia, Drug-Induced; Dyskinesias
Keywords: Parkinson's disease; Dyskinesia; Levodopa-induced Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced; Dyskinesias | interventions — 6-fluoro-2-(4-(pyridin-2-yl)but-3-yn-1-yl)imidazo(1,2-a)pyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dipraglurant TID (Experimental)
  Interventions: Drug: Dipraglurant
- Placebo TID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dipraglurant — Oral 50mg and 100mg tablet
  Other Names: ADX48621
  Arms: Dipraglurant TID
Drug: Placebo — Oral matching placebo tablet
  Arms: Placebo TID

SUMMARY:
This study is designed to evaluate the safety and efficacy of dipraglurant in PD patients with dyskinesia (randomized 1:1 to receive active or placebo) for 12 weeks (1 week at 150 mg per day and 11 weeks at 300 mg per day). The primary efficacy assessment will be based on the Unified Dyskinesia Rating Scale (UDysRS). Patients who complete the 12-week blinded treatment period may have the option to roll into an open-label safety extension study for an additional 12-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease on a stable regimen of antiparkinson's medications, including a levodopa preparation administered not less than 3 times daily.
* Meet protocol-specified criteria for moderate to severe dyskinesia symptoms based on UDysRS and Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) assessments.
* Meet protocol specified criteria for ON time with troublesome dyskinesia based on a standard PD home diary.

Exclusion Criteria:

* Prior surgical treatment for Parkinson's Disease (e.g., deep brain stimulation).
* Other neurological disease (including psychiatric disease and/or cognitive impairment) that, in the opinion of the investigator, would affect the patient's ability to complete study assessments.
* Other significant medical condition that may affect the safety of the patient or preclude adequate participation in the study.
* Pregnant or breast-feeding. Female patients who are of child-bearing potential must be using adequate contraceptive methods (e.g. oral contraceptive, double-barrier method, intra-uterine device, intra-muscular hormonal contraceptive), and have a negative pregnancy test at Screening.

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Unified Dyskinesia Rating Scale (UDysRS) total score | Baseline (Day 1) to Week 12
  The UDysRS is a dyskinesia rating scale scored from 0-104 that evaluates involuntary movements associated with PD. A higher score indicates more severe dyskinesia.

SECONDARY OUTCOMES:
Change from baseline in ON time without troublesome dyskinesia based on a standardized PD diary | Baseline (Day 1) to Week 12
  A PD home diary is used to score 5 different conditions in 30-minute time intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
Change from baseline in OFF time based on a standardized PD diary | Baseline (Day 1) to Week 12
  A PD home diary is used to score 5 different conditions in 30-minute time intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Xenosciences Inc, Phoenix, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - University of California Irvine Medical Center, Irvine, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Pacific Neuroscience Institute, Torrance, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Chase Family Movement Disorders Center - Vernon, Vernon, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton Inc, Boca Raton, Florida
  - Renstar Medical Research -21 NE 1st Ave, Ocala, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - Orlando, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Suncoast Neuroscience Associates Inc, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Geodyssey Research LLC, Vero Beach, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - NeuroStudies.net, LLC - ClinEdge - PPDS, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Josephson Wallack Munshower Neurology PC, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Health System, Bingham Farms, Michigan
  - Michigan State University, East Lansing, Michigan
  - Cooper University Hospital, Camden, New Jersey
  - Rutgers, the State University of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - David L Kreitzman MD PC, Commack, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Toledo, Gardner-McMaster Parkinson Center, Toledo, Ohio
  - Abington Neurologic Associates, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Avera Medical Group, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Health Science Center, San Antonio, San Antonio, Texas
  - Meridian Clinical Research (Norfolk, Virginia), Norfolk, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No